CLINICAL TRIAL: NCT03361514
Title: Discontinuation of Antidepressant Medication in Primary Care Supported by Monitoring Plus Mindfulness-based Cognitive Therapy Versus Monitoring Alone.
Brief Title: Discontinuation of Antidepressant Medication in Primary Care.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Pro Persona Mental Health Care Foundation (Other); Innovatiefonds Zorgverzekeraars (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MFN-ADM-2015-2019; NL56937.091.16 (Registry Identifier: CMO)
Record Dates: First submitted 2017-10-30; First posted 2017-12-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Antidepressants
Keywords: antidepressants, discontinuation, primary care, MBCT
MeSH Terms: interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: This study is designed as a cluster-randomized controlled trial conducted in primary care, randomizing General Practitioners over a.) Supported Protocolized Discontinuation (SPD) alone or b.) SPD with additional Mindfulness-Based Cognitive Therapy (MBCT). Both the patient, GP and the research team will be aware of the allocated condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supported Protocolized Discontinuation (Active Comparator): Supported Protocolized Discontinuation (SPD) Patients will receive guidance of their GP and can have supportive meetings with the mental health assistant.
  Interventions: Behavioral: Supported Protocolized Discontinuation (SPD)
- SPD + Mindfulness (MBCT) (Experimental): In addition to the SPD (as mentioned above) patients are offered Mindfulness Based Cognitive Therapy (MBCT)
  Interventions: Behavioral: Supported Protocolized Discontinuation (SPD); Behavioral: Mindfulness Based Cognitive Therapy (MBCT)

INTERVENTIONS:
Behavioral: Supported Protocolized Discontinuation (SPD) — Patients who choose to discontinue their medication will make a personal tapering schedule with their GP based upon a discontinuation protocol with tapering suggestions. The protocol offers suggestions to taper within a maximum of 6 months describing all types of available dosages per antidepressant so individualized schedules can be constructed. In addition, they will be offered supportive meetings with the GP's mental health assistant. The assistant will receive basic information about discontinuation guidance, i.e. the information brochure, decision aid, discontinuation protocol and a short guideline how to organise consultations.
Behavioral: Mindfulness Based Cognitive Therapy (MBCT) — In addition to the SPD patients are offered Mindfulness Based Cognitive Therapy (MBCT) in homogeneous groups of patients willing to withdraw from their medication. MBCT will be offered according to the treatment protocol developed for recurrent depression, adaptated to the specific needs of patients discontinuing their antidepressant medication. The mindfulness courses will be provided by teachers qualifying the advanced criteria of the Association of Mindfulness Based Teachers in the Netherlands and Flanders. All teachers will receive additional training in using the specific study protocol at the start of the project.
  Arms: SPD + Mindfulness (MBCT)

SUMMARY:
To investigate the effectiveness of the combination of Supported Protocolized Discontinuation (SPD) and Mindfulness-Based Cognitive Therapy (MBCT) in comparison with SPD alone in successful discontinuation of long-term use of antidepressants in primary care.

DETAILED DESCRIPTION:
Antidepressant use continues to rise, mainly explained by an increase in the proportion of patients receiving long term treatment. Although treatment guidelines recommend discontinuation after sustained remission, discontinuing antidepressants appears to be challenging for both patients and general practitioners. Mindfulness-Based Cognitive Therapy (MBCT) is an effective intervention that reduces the risk of relapse in recurrent depression and might facilitate discontinuation by teaching patients to cope with withdrawal symptoms and fear of relapse. The current study aims to investigate the effectiveness of the combination of Supported Protocolized Discontinuation (SPD) and MBCT in comparison with SPD alone in successful discontinuation of long-term use of antidepressants in primary care.

Methods/Design This study involves a cluster-randomized controlled trial conducted in primary care patients with long-term use antidepressants with baseline and 6, 9 and 12 months follow-up assessments. Patients choosing to discontinue their medication will be offered a combination of supported protocolized discontinuation (SPD) and MBCT or SPD alone. Our primary outcome will be full discontinuation of antidepressant medication (= 0 mg) within 6 months after baseline assessment. Secondary outcome measures will be the severity of withdrawal symptoms, symptoms of depression and anxiety, psychological well-being, quality of life and medical and societal costs.

ELIGIBILITY:
Inclusion Criteria:

• Having received prescriptions for antidepressants in primary care for at least the past nine months

Exclusion Criteria:

* Current treatment by a psychiatrist
* Current diagnosis of substance use disorder
* Non-psychiatric indication for long-term antidepressant usage (i.e. neuropathic pain)
* Having participated in a mindfulness training (> 3 sessions) within the last 5 years
* Inability to perform the assessments due to cognitive or language difficulties
* Younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who fully discontinued their antidepressant medication after 6 months. | 6 months
  Our primary outcome will be full discontinuation of antidepressant medication (= 0 mg) within 6 months after baseline assessment. Use of medication will be measured with daily calendars. Patients daily fill out paper calendars describing their daily milligrams of their antidepressant use.

SECONDARY OUTCOMES:
Structured Clinical Interview for DSM-IV-TR Disorders | baseline and 6, 9 and 12 months
  Diagnostic instrument to assess relapse of depressive episode
Discontinuation-Emergent Signs and Symptoms | baseline and 6, 9 and 12 months
  Self-report measure for assessing signs and symptoms associated with discontinuation or interruption of SSRI treatment.
Inventory of Depressive Symptomatology | baseline and 6, 9 and 12 months
  A clinican-administered interview assessing the severity of depressive symptoms
State/Trait Anxiety Inventory | baseline and 6, 9 and 12 months
  Self-report measure for assessing both state and trait levels of anxiety
Module Suicide Cognitions of the Mini International Neuropsychiatric Interview | baseline and 6, 9 and 12 months
  A clinican-administered interview assessing the suicidal cognitions and to specify suicidal risk
Mental Health Continuum - short form | baseline and 6, 9 and 12 months
  Self-report questionnaire that assesses emotional, psychological and social well-being
Five Facet Mindfulness Questionnaire | baseline and 6, 9 and 12 months
  Self-report measure assessing mindfulness skills
Self-Compassion Scale | baseline and 6, 9 and 12 months
  Self-report measure consisting of 12 items addressing six components: self-kindness, self-judgment, common humanity, isolation, mindfulness and over-identification

OTHER OUTCOMES:
Trimbos/iMTA Questionnaire on Costs associated with Psychiatric illness | baseline and 6, 9 and 12 months
  Health service receipt self-report measure designed for economic evaluations in the Netherlands
Euro-Quality of Life 5D-5L | baseline and 6, 9 and 12 months
  Short self-report instrument to assess quality adjusted life years

CONTACTS AND LOCATIONS:
Overall Officials: Anne EM Speckens, prof. dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre for Mindfulness, Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We intend to comply with guidelines for open access as much as possible.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of the main trial papers including embargo period.
Access Criteria: To be decided in a later stage.

REFERENCES:
- [Derived] Huijbers MJ, Wentink C, Lucassen PLBJ, Kramers C, Akkermans R, Spijker J, Speckens AEM. Supporting antidepressant discontinuation using mindfulness plus monitoring versus monitoring alone: A cluster randomized trial in general practice. PLoS One. 2023 Sep 5;18(9):e0290965. doi: 10.1371/journal.pone.0290965. eCollection 2023. PMID 37669281
- [Derived] Wentink C, Huijbers MJ, Lucassen P, Kramers C, Akkermans R, Adang E, Spijker J, Speckens AEM. Discontinuation of antidepressant medication in primary care supported by monitoring plus mindfulness-based cognitive therapy versus monitoring alone: design and protocol of a cluster randomized controlled trial. BMC Fam Pract. 2019 Jul 26;20(1):105. doi: 10.1186/s12875-019-0989-5. PMID 31349796